CLINICAL TRIAL: NCT07117240
Title: Efficacy of Treatment Strategies for Steroid-induced Diabetes - a Comparison of GLP-1 Receptor Agonist Plus Basal Insulin With Intensive Insulin Therapy
Brief Title: Evaluation of the Efficacy and Safety of GLP-1 Receptor Agonist Therapy In Steroid-Induced Diabetes
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Aleksandra Jedrasek, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KB/113/2025
Record Dates: First submitted 2025-07-28; First posted 2025-08-12 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Steroid-Induced Diabetes; Steroid-Induced Hyperglycemia; Diabetes
Keywords: Steroid-induced diabetes; GLP-1 receptor agonist; Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — lixisenatide; Insulin Glargine; Glucagon-Like Peptide 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with Steroid-Induced Diabetes (Experimental): Patients diagnosed with Steroid-induced diabetes, that require insulin therapy
  Interventions: Drug: lixisenatide + glargine; Drug: Intensive insulin therapy
- Patients with type 2 diabetes and Steroid-Induced Hyperglycaemia (Experimental): Patients with history of type 2 diabetes, that developed Steroid-induced hyperglycaemia and require insulin therapy
  Interventions: Drug: lixisenatide + glargine; Drug: Intensive insulin therapy

INTERVENTIONS:
Drug: lixisenatide + glargine — Participants assigned to Group 1 will receive standard insulin therapy. Those in Group 2 will be treated with a combination of insulin glargine and lixisenatide, with dosages individually adjusted based on current glucose levels. All participants will be trained in insulin administration and dose adjustment based on glucose readings.
  Other Names: GLP-1 plus basal insulin
Drug: Intensive insulin therapy — Participants assigned to Group 1 will receive standard insulin therapy. Those in Group 2 will be treated with a combination of insulin glargine and lixisenatide, with dosages individually adjusted based on current glucose levels. All participants will be trained in insulin administration and dose adjustment based on glucose readings.

SUMMARY:
Glucocorticoids are commonly used in the treatment of autoimmune, inflammatory, and neoplastic diseases. Despite their therapeutic efficacy, they are associated with significant metabolic side effects. In the proposed research, the aim is to assess the metabolic efficacy and safety of fixed-ratio combination therapy (basal insulin + GLP-1 receptor agonist) compared to standard insulin therapy in patients with SID. In a selected group of patients, a randomised clinical trial would be conducted to assess the potential benefits of GLP-1 receptor agonists in the management of SID.

DETAILED DESCRIPTION:
Glucocorticoids are commonly used in the treatment of autoimmune, inflammatory, and neoplastic diseases. Despite their therapeutic efficacy, they are associated with significant metabolic side effects. Their strongly diabetogenic effect results from the enhanced activity of hyperglycemic hormones, increased insulin resistance, and impaired function of pancreatic β-cells. Current clinical guidelines classify SID as a form of drug-induced diabetes, with insulin therapy as the primary treatment. However, recent studies highlight the role of glucocorticoids in exacerbating insulin resistance, inhibiting incretin effects, and promoting weight gain-factors that suggest a potential therapeutic role for GLP-1 receptor agonists. It is estimated that approximately 100 patients will be needed to achieve statistically significant results. Participants will be stratified based on the type of diabetes (type 2 diabetes vs. steroid-induced diabetes), followed by alternate randomisation into one of two therapeutic groups:

Group 1: Patients receiving insulin therapy Group 2: Patients receiving an FRC therapy (insulin glargine and lixisenatide) A clinical research team will perform body composition analysis using bioelectrical impedance analysis (BIA) with a Tanita scale. To assess baseline metabolic control, blood samples will be taken. All study participants will be equipped with a CGM sensor integrated with the hospital clinic system, allowing the study team access to the patients' glycemic data.

Participants assigned to Group 1 will receive standard insulin therapy. Those in Group 2 will be treated with a combination of insulin glargine and lixisenatide, with dosages individually adjusted based on current glucose levels. All participants will be trained in insulin administration and dose adjustment based on glucose readings. After hospital discharge, patients will continue to be monitored by the study team using data from the CGM system. The researcher will frequently assess the Glucose Management Indicator (GMI), Time in Range (TIR), daily insulin requirements, and frequency of hypoglycemic episodes.

Follow-up phone calls will be attempted every 2 months. If two consecutive contact attempts are unsuccessful, the study will continue based solely on CGM data. A final follow-up visit will take place after 6 months. During this visit, body composition will be reassessed, and the Diabetes Treatment Satisfaction Questionnaire (DTSQ) will be administered to evaluate patient-reported quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years of age)
* Patients with type 2 diabetes and SIH, or diagnosed with SID requiring insulin
* Patients undergoing long-term oral GC therapy for the following indications:
* Nephrotic syndrome
* Asthma
* Rheumatoid arthritis
* Psoriatic arthritis
* Polymyalgia rheumatica
* Synovitis associated with osteoarthritis
* Sarcoidosis
* Tubulointerstitial nephritis
* Atopic dermatitis
* Pemphigus
* Informed consent

Exclusion Criteria:

* - Age <18 years
* Type 1 diabetes
* Critically ill patients in a life-threatening condition requiring intensive care and medical support to sustain vital functions, as defined by an Allgöwer index >1.0
* eGFR <30 mL/min
* History of acute pancreatitis or gallstone disease
* Lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2028-02-09 (Estimated); Study Completion 2028-07-10 (Estimated)

PRIMARY OUTCOMES:
Glucose monitoring index and Time in range | From enrollment to 6 months
  Achievement of glycemic targets measured through Continuous Glucose Monitoring Sensor. Glycemic goals were established at:
  GMI ≤ 7.0% TIR > 70% (glucose 70-180 mg/dL)

SECONDARY OUTCOMES:
Need for prandial insulin in Group 2 (glucose >200 mg/dL in ≥2 measurements over 2 days) | From enrollment to 6 months
Assessment of body mass index (BMI) | Measurements will be taken at the time of enrollment and again after 6 months
  weight and height will be combined to report BMI in kg/m^2
Patient satisfaction assessed using the Diabetes Treatment Satisfaction Questionnaire | From enrollment to 6 months
  Treatment Satisfaction is rated between 0 and +18, the higher the score the greater the satisfaction with treatment.
Number of patients that refused to initiate therapy or discontinued therapy due to personal and/or financial reasons | From enrollment to 6 months
  The number of patients that refused to initiate or continue therapy will be measured based on patient's declaration and monthly evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Leszek Czupryniak, Prof. Dr. hab.n.med., Study Director — Medical University of Warsaw
Locations (1):
- Warsaw Medical University, Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No